CLINICAL TRIAL: NCT06651606
Title: Using Behavioral Economics to Mitigate Relapse of Problem Behavior in an Intellectual and Developmental Disabilities Population
Brief Title: Preventing Relapse of Problem Behavior Through Behavioral Economics: A Translational Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Collaborators: Auburn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD113794-01A1 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Problem Behavior
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive Ratio Training (Experimental): Participants in the progressive ratio training Arm will experience the novel reinstatement-mitigation tactic: Progressive Ratio Training (PRT).
  Progressive ratio training (PRT) is used to prevent recurrence of the proxy response when extinction errors occur. PRT involves providing a reinforcer for the proxy response on a geometric progressive ratio (PR) scale. The schedule requirement will increase for the target response each time a reinforcer is delivered. For example, once a reinforcer is delivered on the PR-2 schedule, the requirement will increase to a PR-4, then to a PR-8, -16,
  -32, etc.
  Interventions: Behavioral: Progressive Ratio Training (PRT)
- Standard of Care (Experimental): Participants in the standard of care Arm will receive an analogue to the standard of care approach for problem behavior: differential reinforcement of alternative behavior (DRA) with extinction.
  In DRA with extinction, the proxy for problem behavior will cease to produce reinforcement while the proxy for communication behavior will produce reinforcement on a fixed-ratio 1 schedule of reinforcement.
  Interventions: Behavioral: Differential Reinforcement of Alternative (DRA) Behavior with Extinction

INTERVENTIONS:
Behavioral: Progressive Ratio Training (PRT) — Progressive ratio training (PRT) is used to prevent recurrence of the proxy response when extinction errors occur. PRT involves providing a reinforcer for the proxy response on a geometric progressive ratio (PR) scale. The schedule requirement will increase for the target response each time a reinforcer is delivered. For example, once a reinforcer is delivered on the PR-2 schedule, the requirement will increase to a PR-4, then to a PR-8, -16,
  -32, etc.
  Arms: Progressive Ratio Training
Behavioral: Differential Reinforcement of Alternative (DRA) Behavior with Extinction — In DRA with extinction, the proxy for problem behavior is placed on extinction and no longer produces reinforcement. The proxy for communication behavior produces reinforcement on a fixed-ratio 1 schedule of reinforcement.
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to compare a novel tactic for mitigating reinstatement compared to the current standard of care approach using a translational-treatment model. The main questions it aims to answer are:

1. how well does progressive ratio training mitigate response-dependent reinstatement compared to the standard of care approach?
2. how well does progressive ratio training mitigate response-independent reinstatement compared to the standard of care approach?

DETAILED DESCRIPTION:
Behavioral treatments can be an effective means to treat problem behavior. One of the most common behavioral treatments is differential reinforcement of alternative behavior, frequently implemented as functional communication training. Most demonstrations of behavioral treatments, including functional communication training, are conducted in highly controlled settings by trained therapists. When these treatments are implemented in community settings (e.g., an individual's home) by caregivers, they will be challenged, which can lead to the recurrence and sustained relapse of problem behavior. Recurrence and relapse can be the first step in a chain that leads to treatment failure. Fortunately, some tactics have been designed to sustain treatment effectiveness and mitigate two forms of relapse (i.e., resurgence and renewal) that result from two of three primary treatment challenges. These tactics function as inoculation (i.e., make problem behavior less likely to return). However, there are no tactics designed to specifically mitigate a third form of relapse: reinstatement

This project involves a novel inoculation tactic to mitigate reinstatement and protect against the third common treatment challenge: extinction errors. The tactic in question is based on substantial conceptual and empirical evidence from behavioral economics, as well as the investigators' pilot work. The project uses an innovative translational-treatment model to better understand which of the proposed tactics (our novel tactic or the default standard-of-care approach) better inoculates against extinction errors through real-world analogues. The use of a translational-treatment model is consistent with other research examining the role of basic processes in behavioral treatment when collateral effects are unknown, and will also engender a thorough examination of the proposed tactics.

In Aim 1, investigators will establish a proxy response, apply treatment to that proxy response, and examine the effectiveness of progressive ratio training in inoculating against extinction errors and mitigating response-dependent reinstatement.

In Aim 2, investigators will establish a proxy response, apply treatment to that proxy response, and examine the effectiveness of progressive ratio training in inoculating against extinction errors and mitigating response-independent reinstatement. Outcomes of this research could improve the current standard of care for behavioral treatments to make them more effective in community application, result in the development and validation of novel inoculation tactics, and significantly improve the lives of individuals with IDD.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls from ages 6 to 21
* Engage in problem behavior
* Diagnosis of some type of intellectual and developmental disability

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Treatment Effectiveness | 2 years
  The number of individuals for whom treatment remains effective (either progressive ratio training or current standard-of-care), which investigators will determine by comparing the mean rate of responding in baseline and subsequent conditions (Treatment and Reinstatement Tests 1 and 2). If investigators find at least an 80% reduction in target behavior in a condition (a standard clinical target for problem behavior), they will conclude that the treatment is effective (or remains effective).

SECONDARY OUTCOMES:
Proportional and Comparative Effectiveness | 2 years
  The proportional and comparative effectiveness of the treatments, which investigators will determine from the mean rate of behavior in Phase 2 Treatment and the treatments during Phase 3 Reinstatement Tests (with progressive-ratio training and the standard-of-care approach), and determine the difference in percent reduction between treatment and the reinstatement tests. This second measure is preliminary: no pilot data speak to what may be observed. However, these data are likely to be important to future research.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Kranak, PhD, Principal Investigator — Oakland University
Locations (2):
- United States (2):
  - Auburn University, Auburn, Alabama
  - Oakland University, Rochester, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share outcome data as specified in the approved Data Management and Sharing Plan.
Time Frame: Data will become available at the completion of the study as specified in the approved Data Management and Sharing Plan.
Access Criteria: Data will be accessible as specified in the approved Data Management and Sharing Plan.